CLINICAL TRIAL: NCT06369675
Title: A 21-Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of MOB015B in Healthy Subjects Using a Cumulative Irritant Patch Test Design
Brief Title: Skin Irritation Potential of MOB015B in Healthy Subjects Using a Cumulative Irritant Patch Test Design
Acronym: CIPT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MOB015B-V
Record Dates: First submitted 2017-08-01; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Erythema
MeSH Terms: conditions — Erythema | interventions — long-chain-aldehyde dehydrogenase; Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MOB015B, MOB015B vehicle, 0.2% SLS and an inert control (Experimental): All subjects will receive MOB015B, MOB015B vehicle, 0.2% SLS (positive control) and inert control (negative control) Each subject will serve as his or her own control
  Interventions: Drug: MOB015B; Drug: 0.2% SLS; Drug: 0.9% Saline; Drug: MOB015B vehicle

INTERVENTIONS:
Drug: MOB015B — Topical formulation
Drug: 0.2% SLS — Positive control
Drug: 0.9% Saline — Negative control
Drug: MOB015B vehicle — Topical formulation

SUMMARY:
A 21-Day, Randomized, Controlled Study to Evaluate the Skin Irritation Potential of MOB015B in Healthy Subjects Using a Cumulative Irritant Patch Test Design To evaluate the irritation potential of MOB015B on normal skin. Single center, randomized, controlled, evaluator blinded, within-subject comparison study

DETAILED DESCRIPTION:
MOB015B is a newly developed topical solution for the treatment of nail fungus (onychomycosis) containing the active antifungal ingredient terbinafine. A This study investigates the irritation potential of MOB015B under standardized conditions compared with a known irritant (0.2% SLS) and an inert control (normal saline). Because MOB015B is formulated for topical use, it is necessary to determine the potential of this product to cause irritation after repeated topical application to the skin.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible for participation in the study if all of the following inclusion criteria are satisfied prior to randomization:

1. Is a healthy male or female (to be confirmed by medical history);
2. Is 18 years of age or older;
3. In the case of a female of childbearing potential, is using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy, tubal ligation). Abstinence or vasectomies are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
4. In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) on Day 1 prior to randomization and are willing to submit to a UPT at the end of study (EOS);
5. Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs;
6. Is of any Fitzpatrick Skin Type or race, providing the skin pigmentation will allow discernment of erythema
7. Complete a medical screening procedure; and
8. Read, understand, and sign an informed consent.

Exclusion Criteria:

1. Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction;
2. Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
3. Is not willing to refrain from using systemic/topical anti-inflammatory analgesics such as aspirin (81 mg daily aspirin will be allowed), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
4. Is using medication which, in the opinion of the Investigator, will interfere with the study results (e.g. anti-inflammatory medications, antipsychotics, anticonvulsants with potential pain relief effects, immunomodulatory medications, and others);
5. Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study;
6. Has psoriasis and/or active atopic dermatitis/eczema;
7. Has a known sensitivity or allergy to constituents of the materials being evaluated;
8. Is a female who is pregnant, plan to become pregnant during the study, or is breast feeding a child;
9. Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
10. Has received treatment for any type of internal cancer within 5 years prior to study entry;
11. Has a history of, or are currently being treated for skin cancer and/or hepatitis;
12. Has a history of, or is currently being treated for, insulin dependent diabetes;
13. Has any condition that might compromise study results;
14. Currently or expect to sunbathe or use tanning salons during the study;
15. Is currently participating in any clinical testing;
16. Has any known sensitivity to adhesives; and/or
17. Has received any investigational drug(s) within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
To determine the potential of MOB015B to cause skin irritation after repeated topical application to the healthy skin of humans under controlled conditions. | 22 days
  The mean cumulative irritation score
To assess safety | 22 days
  Safety was assessed by evaluation of any AEs reported during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Dosik, MD, Principal Investigator — TKL Research
Locations (1):
- TKL Research, Inc, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No